CLINICAL TRIAL: NCT05965648
Title: Families FORWARD: Development of a Family-Based Transition Planning Program for Culturally-Diverse Youth on the Autism Spectrum
Brief Title: Development of a Family-Based Transition Planning Program for Culturally-Diverse Youth on the Autism Spectrum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Deborah Munroe Noonan Memorial Research Fund (Other)
Responsible Party: Principal Investigator, Kristin Long, Associate Professor, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6444E
Record Dates: First submitted 2023-06-28; First posted 2023-07-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder; Family Relations
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Families FORWARD (Other): This is a single-arm trial of a new transition planning program for families of youth on the autism spectrum. The program includes six or seven bi-weekly parent sessions, three of which are optional for the youth to attend. The program will be facilitated by community-based service providers who work with transition-aged youth on the autism spectrum and/or their families.
  Interventions: Behavioral: Families FORWARD (Focusing on Relationships, Well-being, and Responsibility aheaD)

INTERVENTIONS:
Behavioral: Families FORWARD (Focusing on Relationships, Well-being, and Responsibility aheaD) — Families FORWARD aims to engage families in planning for adulthood earlier and more actively. Program skills include communication and problem-solving; guided practice in setting realistic goals, breaking down goals into incremental action steps, and problem-solving barriers to goal attainment; repeated engagement in future-oriented communication; and training on how to navigate transition-related and adult services. Parents/caregivers will participate in six or seven telehealth sessions (60-75 minutes each). Youth on the autism spectrum will have the option of participating in up to three program sessions to increase collaborative planning within the family. Families will identify and work toward individualized transition planning goals that may fall within any area of planning or functioning (e.g., housing, education, guardianship).

SUMMARY:
The goal of this clinical study is to develop a community-based program to support family members of transition-aged youth on the autism spectrum to help them plan for the future. The main aims of the study are:

1. To develop the Families FORWARD program
2. To conduct proof-of-concept testing of the Families FORWARD program

Participants will complete surveys before and after participating in the program and will participate in exit interviews at the end of the program.

DETAILED DESCRIPTION:
The Families FORWARD (Focusing on Relationships, Well-being, and Responsibility aheaD) program aims to increase family members' active planning for the transition to adulthood in the context of autism. The program is designed to enable flexible delivery for families of youth who are diverse across autism features, co-occurring conditions, service needs, cultural values and preferences, and readiness to engage in planning. The program will be delivered collaboratively with community organizations that support individuals on the autism spectrum and/or their families.

The current project aims to conduct proof-of-concept testing with a culturally-diverse sample of families of transition-aged youth on the autism spectrum. Parents / primary caregivers will participate in 6-7 individual, personalized sessions that incorporate aspects of skill-building (communication, goal-setting, problem-solving, systems navigation), education about services, and motivational interviewing. Youth will be invited to participate in 3 of the sessions along with their parent / primary caregiver. Participants will complete surveys before and after participating in the program and will participate in exit interviews at the end of the program. The investigators will assess indicators of acceptability, feasibility, and improvement on proposed mediators and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Family Inclusion Criteria

  1. Parents or primary caregivers of transition-aged youth on the autism spectrum:

     1. Have one or more child(ren) on the autism spectrum who is/are ages 14-21 years old
     2. Identify as the parent, legal guardian, and/or primary caregiver of the youth
     3. Speak English fluently
     4. Reside in Massachusetts
  2. Youth on the autism spectrum:

     1. Have an autism diagnosis OR identify as autistic
     2. Age 14-21
     3. Have ability to communicate verbally or in written format in English
     4. Reside in Massachusetts

Exclusion Criteria: none

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Families FORWARD Program Acceptability Form | At the conclusion of all sessions in the program (approximately 3 months)
  The parents (and youth, when applicable) will complete the Program Acceptability scale that will assess acceptability, appropriateness, and feasibility. Item scores range from 0 to 4. Higher scores are associated with higher perceptions of intervention acceptability, appropriateness, and feasibility.
Transition Planning Activities | Baseline, 3 months
  The Transition Planning Activity Measure will be used to assess parent's readiness for their youth's transition to adulthood. It is a parent proxy questionnaire. Item scores range from 1 to 4. Higher scores are associated with higher transition readiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.